CLINICAL TRIAL: NCT06202651
Title: Treatment of Granular Corneal Dystrophy Using Nd-YAG Laser
Brief Title: Neodymium-doped Yttrium Aluminum Garnet (Nd:YAG) Laser Treatment for Granular Corneal Dystrophy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was no change in size of the Nd:YAG laser-treated GCD deposits as assessed by the various modalities on visit 2, and it was decided to terminate the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00304623
Record Dates: First submitted 2023-12-23; First posted 2024-01-11 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Granular Dystrophy, Corneal
Keywords: Granular Dystrophy; Cornea; Nd:YAG Laser; Neodymium-doped Yttrium Aluminum Garnet Laser
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: A single interventional group of Granular Corneal Dystrophy participants over the age of 18 years that undergo a single Neodymium-doped Yttrium Aluminum Garnet (Nd:YAG) Laser treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nd:YAG Laser Interventional Cohort (Experimental): Participants include Granular Corneal Dystrophy patients.
  On visit 1, participants will undergo visual acuity testing, slit-lamp examination, intra-ocular pressure (IOP) measurement, Scheimpflug tomography, anterior-segment optical coherence tomography (AS-OCT), and slit-lamp photography of the cornea.
  On the same visit or on a separate visit within 1 month, the participants will undergo the Nd:YAG Laser treatment. At the investigators' discretion, after the procedure, participants might need to administer generic topical antibiotic eye drops three times daily for a week.
  One week post-intervention (visit 2), the participant will repeat visual acuity testing, slit-lamp examination, IOP measurement, Scheimpflug tomography, AS-OCT, and slit-lamp photography of the cornea.
  Three months post-intervention (visit 3), the participant will repeat visual acuity testing, slit-lamp examination, IOP measurement, Scheimpflug tomography, AS-OCT, and slit-lamp photography of the cornea.
  Interventions: Device: Nd:YAG Laser

INTERVENTIONS:
Device: Nd:YAG Laser — Prior to Nd:YAG laser treatment, two drops of topical anesthetic will be administered to the study eye. The two most peripheral deposits that are of ca. 50 µm size will be located and used as the targets for the treatment. The Nd:YAG laser will then be administered to each one of the two deposits, beginning with the lowest energy setting (0.3 mJ) and increasing the energy levels up to to 3 mJ in increments of 0.5 mJ. Five single-burst shots will be performed per laser energy setting per opacity until a visible effect is seen.
  After the procedure, the eye will be examined to assess the integrity of the corneal epithelium. If a defect is seen, the participant will be advised to administer topical antibiotic eye drops three times daily for a week as a precautionary measure.
  Other Names: Optimis II (Quantel Medical)

SUMMARY:
Granular Corneal Dystrophy is a rare hereditary disease characterized by the development of deposits within the cornea, which may in turn affect the quality of vision. Still today, all existing treatment options are based on surgical intervention and there is no minimally-invasive treatment available for the disease.

The goal of this clinical trial is to test the effectiveness and safety of Neodymium-doped yttrium aluminum garnet (Nd:YAG) laser as a minimally-invasive treatment for people suffering from Granular Corneal Dystrophy. The main question it aims to answer is if Nd:YAG laser is able to disintegrate the characteristic corneal depositions in a safe manner without causing significant adverse effects.

If found suitable to be part of the study, participants will first undergo a series of imaging studies to measure and characterize the corneal deposits. After completion, the participants will undergo the Nd:YAG laser treatment under local anesthesia by a corneal specialist, targeting deposits not involving the visual axis. Following the treatment, participants might need to take antibiotic eye drops for a duration of approximately one week. The participants will be required to attend two follow-up visits: one week after the treatment and 3 months after the treatment. In each one of the follow-up visits, an eye examination will be performed and the same series of imaging studies that was performed prior to the Nd:YAG laser treatment will be repeated.

DETAILED DESCRIPTION:
Neodymium:yttrium aluminum garnet (Nd:YAG) laser is an ophthalmic instrument that finds versatile use in clinical practice since its first introduction in 1980s. This solid-state laser emits infrared light at a wavelength of 1064 nm that can disrupt ocular tissues by causing an optical breakdown with a short, high-power pulse. Thanks to its high precision, minimal-invasive mode of delivery, and well-established safety profile, its application ranges from treatment of posterior capsule opacification, chronic and acute angle-closure glaucoma, vitreous floaters, to proliferative diabetic retinopathy.

Granular corneal dystrophy (GCD) is a rare hereditary condition characterized by progressive deposition of insoluble protein aggregates in the cornea. The small, white-greyish granular deposits typically begin to form during childhood and grow in size and number with increasing age, eventually coalescing and causing significant visual impairment.

Still today, there is no minimal-invasive treatment available for GCD patients. Current treatment approaches include partial or full-thickness corneal transplant, which is associated with a relatively high recurrence rate and potentially sight-threatening complications. In addition, there is a global shortage of available donor corneas. Therefore, there is an unmet need for a minimal-invasive treatment that could reduce this indication for corneal transplantation and provide symptomatic relief to GCD patients.

As modern Nd:YAG laser systems can focus on a spot size as small as 8-10 µm in different depths of the cornea, the study team hypothesize that the Nd:YAG laser would be capable of accurately targeting the GCD deposits and serve as a viable minimal-invasive treatment option for this disease.

Hence, in the proposed research, the investigators seek to evaluate the efficacy and safety of the Nd:YAG laser in the treatment of GCD patients. If found to be efficacious and safe, the investigators hypothesize that GCD patients will benefit from both the minimal-invasive form of treatment and prompt improvement in quality of life and vision.

During the study, as part of the initial assessment, the participants will undergo routine ophthalmic examination including visual acuity testing, slit-lamp examination, intra-ocular pressure measurement, and corneal imaging including Scheimpflug tomography (Pentacam®), anterior-segment optical coherence tomography (AS-OCT), and slit-lamp photography of the cornea (visit 1). All the above imaging modalities are non-contact, take seconds to perform, and represent no risk to the participant.

Following the initial assessment, the Nd:YAG laser procedure will be performed on the same day (visit 1) or on a separate date (visit 2) depending on the time schedule of both the participant and the research team. One eye will be included in the study per participant. If the severity of the disease is asymmetrical, the eye with more extensive corneal deposition will be included. If the severity is symmetrical, the participant's non-dominant eye will be included as determined by the standard dominance testing method.

Using the slit-lamp, the primary investigator, a corneal specialist, will find the two most peripheral deposits that are of ca. 50 µm size. The width of the thinnest slit-lamp beam, which is 1 mm, will be used as a guide to estimate the deposits' size. The exact size of each opacity will be measured using the images taken by the AS-OCT and slit-lamp photography.

Prior to the Nd:YAG laser treatment, two drops of topical anesthetic will be administered to the study eye to anesthetize the eye, as is always done prior to any other Nd:YAG procedure. The treatment will be delivered using an Optimis II device (Quantel Medical). This is an FDA-approved device used regularly for other ocular indications, that due to its adherence to Non-Significant Risk (NSR) criteria, received an abbreviated Investigational Device Exemption (IDE) approval by the institutional review board (IRB) for the purpose of this study. Typically, a single-pulse Nd:YAG laser energy levels of 2-3 mJ is sufficient to treat posterior capsule opacification, while 2-8 mJ of energy is used to perform an iridotomy. In this research, the primary investigator will begin with the lowest energy setting (0.3 mJ) and increase the energy levels to 3 mJ in increments of 0.5 mJ. Five single-burst shots will be performed per laser energy setting per opacity until a visible effect is seen.

After the procedure, the eye will be examined to assess the integrity of the corneal epithelium. If a defect is seen, the participant will be advised to administer topical antibiotic eye drops three times daily for a week as a precautionary measure. The investigators hypothesize minor risks of corneal scarring or intraocular inflammation after the laser treatment. The participants' visual acuity should not be affected as only peripheral deposits that lie outside the visual axis will be subjected to treatment in this research.

The participant will return one week (visit 2 or 3) and three months (visit 3 or 4) later for follow-up at which the participant will repeat the clinical examination and imaging studies included above. The study cornea will be examined carefully for any signs of inflammation or scarring. The size of the opacities that were treated with Nd:YAG laser will be re-measured using the images taken by the anterior-segment OCT and slit-lamp photography. After the last follow-up examination, the participants will be referred to routine care.

During the entire course of the study, confidentiality will be ensured using standard procedures including storage of study data on password protected computers utilizing a Secure Analytic Framework Environment (SAFE) desktop. Participants will be assigned study identification codes that will be used for all subsequent study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Diagnosis of granular corneal dystrophy with presence of granular opacities in the peripheral cornea of appropriate size (ca. 50 µm) in at least one eye
* Willingness and ability to give signed informed consent and follow study instructions

Exclusion Criteria:

* Presence of any active intra-ocular inflammation
* Pre-existing glaucoma or retinal edema
* Cannot properly self-administer or receive an eye drop medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Change in size of granular corneal deposits due to Nd:YAG laser treatment | Baseline, Post-intervention day 7, Post-intervention 3 months
  The size of each one of the two treated corneal deposits per participant will be measured in µm on images taken by both the AS-OCT and slit-lamp photography in each study visit. The size will be measured both manually and automatically on each one of the imaging techniques. A comparison of the size between study visits will be performed, change from day 7 post-intervention to month 3 post-intervention.

SECONDARY OUTCOMES:
Safety as the number participants experiencing adverse events of inflammation and/or scarring | Post-intervention day 7, Post-intervention 3 months
  Number of participants who experience adverse events of inflammation and scarring after Nd:YAG laser intervention. Inflammation will be defined as grade>1 of cells, flare and/or endothelitis on the visit of day 7 and grade>0 cells, flare and/or endothelitis on the visit of month 3, as defined by the Standardization of Uveitis Nomenclature (SUN) criteria. Any scarring will be considered an adverse event and will be measured in µm by slit-lamp photography and AS-OCT in each follow-up visit.
Safety as the number of participants experiencing decrease in visual acuity | Baseline, Post-intervention day 7, Post-intervention 3 months
  Visual acuity will be tested at baseline and on each follow-up visit. The number of patients who experience a decrease of more than 0.1 LogMAR in visual acuity after the treatment and the amount of decrease in LogMAR will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Albert S Jun, MD, PhD, Principal Investigator — Wilmer Eye Institute/Johns Hopkins University
Locations (1):
- Wilmer Eye Institute - Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Aron-Rosa D. Use of a pulsed neodymium-Yag laser for anterior capsulotomy before extracapsular cataract extraction. J Am Intraocul Implant Soc. 1981 Fall;7(4):332-3. doi: 10.1016/s0146-2776(81)80029-8. No abstract available. PMID 7349647
- [Background] Fankhauser F, Lortscher H, van der Zypen E. Clinical studies on high and low power laser radiation upon some structures of the anterior and posterior segments of the eye. Experiences in the treatment of some pathological conditions of the anterior and posterior segments of the human eye by means of a Nd:YAG laser, driven at various power levels. Int Ophthalmol. 1982 May;5(1):15-32. doi: 10.1007/BF00129992. PMID 7118438
- [Background] Vogel A, Busch S, Jungnickel K, Birngruber R. Mechanisms of intraocular photodisruption with picosecond and nanosecond laser pulses. Lasers Surg Med. 1994;15(1):32-43. doi: 10.1002/lsm.1900150106. PMID 7997046
- [Background] Jagger JD. The Nd-YAG Laser in Ophthalmology: Principles and Clinical Applications of Photodisruption. Br J Ophthalmol. 1986;70(1):79.
- [Background] Blumenkranz MS. The evolution of laser therapy in ophthalmology: a perspective on the interactions between photons, patients, physicians, and physicists: the LXX Edward Jackson Memorial Lecture. Am J Ophthalmol. 2014 Jul;158(1):12-25.e1. doi: 10.1016/j.ajo.2014.03.013. Epub 2014 Mar 31. PMID 24699157
- [Background] Ficker LA, Steele AD. Complications of Nd:YAG laser posterior capsulotomy. Trans Ophthalmol Soc U K (1962). 1985;104 ( Pt 5):529-32. PMID 3863341
- [Background] Karahan E, Er D, Kaynak S. An Overview of Nd:YAG Laser Capsulotomy. Med Hypothesis Discov Innov Ophthalmol. 2014 Summer;3(2):45-50. PMID 25738159
- [Background] Munier FL, Frueh BE, Othenin-Girard P, Uffer S, Cousin P, Wang MX, Heon E, Black GC, Blasi MA, Balestrazzi E, Lorenz B, Escoto R, Barraquer R, Hoeltzenbein M, Gloor B, Fossarello M, Singh AD, Arsenijevic Y, Zografos L, Schorderet DF. BIGH3 mutation spectrum in corneal dystrophies. Invest Ophthalmol Vis Sci. 2002 Apr;43(4):949-54. PMID 11923233
- [Background] Weiss JS, Moller HU, Aldave AJ, Seitz B, Bredrup C, Kivela T, Munier FL, Rapuano CJ, Nischal KK, Kim EK, Sutphin J, Busin M, Labbe A, Kenyon KR, Kinoshita S, Lisch W. IC3D classification of corneal dystrophies--edition 2. Cornea. 2015 Feb;34(2):117-59. doi: 10.1097/ICO.0000000000000307. PMID 25564336
- [Background] Ellies P, Renard G, Valleix S, Boelle PY, Dighiero P. Clinical outcome of eight BIGH3-linked corneal dystrophies. Ophthalmology. 2002 Apr;109(4):793-7. doi: 10.1016/s0161-6420(01)01025-9. PMID 11927442
- [Background] Seitz B, Behrens A, Fischer M, Langenbucher A, Naumann GO. Morphometric analysis of deposits in granular and lattice corneal dystrophy: histopathologic implications for phototherapeutic keratectomy. Cornea. 2004 May;23(4):380-5. doi: 10.1097/00003226-200405000-00013. PMID 15097134
- [Background] Lopes-Ferreira D, Neves H, Queiros A, Faria-Ribeiro M, Peixoto-de-Matos SC, Gonzalez-Meijome JM. Ocular dominance and visual function testing. Biomed Res Int. 2013;2013:238943. doi: 10.1155/2013/238943. Epub 2013 Nov 11. PMID 24319677
- [Background] Bhargava R, Kumar P, Prakash A, Chaudhary KP. Estimation of mean ND: Yag laser capsulotomy energy levels for membranous and fibrous posterior capsular opacification. Nepal J Ophthalmol. 2012 Jan-Jun;4(1):108-13. doi: 10.3126/nepjoph.v4i1.5861. PMID 22344007
- [Background] Drake MV. Neodymium:YAG laser iridotomy. Surv Ophthalmol. 1987 Nov-Dec;32(3):171-7. doi: 10.1016/0039-6257(87)90092-0. PMID 3328316